CLINICAL TRIAL: NCT00003313
Title: A Phase III Randomized Study of Amifostine Mucosal Protection for Patients With Favorable Performance Inoperable Stage II-III A/B Non-Small Cell Lung Cancer (NSCLC) Receiving Sequential Induction and Concurrent Hyperfractionated Radiotherapy With Paclitaxel and Carboplatin
Brief Title: Amifostine in Treating Patients With Stage II or Stage III Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RTOG-9801; CDR0000066260
Record Dates: First submitted 1999-11-01; First posted 2003-11-26 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Drug/Agent Toxicity by Tissue/Organ; Lung Cancer; Oral Complications; Radiation Toxicity
Keywords: stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; oral complications; drug/agent toxicity by tissue/organ; radiation toxicity
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Lung Neoplasms; Radiation Injuries; Carcinoma, Non-Small-Cell Lung | interventions — Filgrastim; Amifostine; Carboplatin; Paclitaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Radiation therapy and chemotherapy + Amifostine
  Interventions: Biological: filgrastim; Drug: amifostine trihydrate; Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy
- Arm 2 (Active Comparator): Radiation therapy and chemotherapy alone
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
  Arms: Arm 1
Drug: carboplatin
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Amifostine may be an effective treatment for the toxic side effects caused by radiation therapy and chemotherapy. It is not yet known whether chemotherapy and radiation therapy are more effective with or without amifostine for non-small cell lung cancer.

PURPOSE: Randomized phase III trial to determine the effectiveness of amifostine in treating patients who have stage II or stage III non-small cell lung cancer that cannot be surgically removed and who are undergoing chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate whether the addition of the radioprotector amifostine can reduce the incidence and severity of non-hematologic toxicity, specifically esophagitis and pneumonitis, during concurrent hyperfractionated radiotherapy and chemotherapy (with paclitaxel and carboplatin) in patients with stage II, IIIA, or IIIB non-small cell lung cancer. II. Evaluate the differences in quality of life and symptom distress, specifically dysphagia, between patients receiving amifostine and those not receiving amifostine. III. Evaluate the relationship of tobacco use and alcohol use during treatment to appraisals of quality of life and symptom distress, specifically esophagitis, in the two groups. IV. Evaluate the efficacy of induction therapy with paclitaxel and carboplatin followed by concurrent chemotherapy and hyperfractionated radiotherapy in these patients.

OUTLINE: This is an open-label treatment and randomized supportive care study. Patients are stratified according to disease stage (II vs IIIA vs IIIB), Karnofsky performance status (90-100% vs 70-80%), and age (70 and under vs over 70). Patients are randomized to one of two treatment arms. Arm I: Patients receive paclitaxel IV over 3 hours on days 1 and 22 and over 1 hour weekly for 6 weeks beginning on day 43. Patients receive carboplatin IV over 30 minutes immediately after each paclitaxel dose. Patients receive filgrastim (G-CSF) subcutaneously for 10-14 days after each of the first two paclitaxel and carboplatin doses. Radiotherapy begins on day 43 and is administered twice daily for 5 days per week for 6 weeks. Beginning on day 43, patients receive amifostine IV over 5-7 minutes 4 days a week for 6 weeks. Arm II: Patients receive treatment as in arm I without amifostine. Quality of life is assessed at baseline, before chemoradiation (after 2 courses of induction chemotherapy), the last week of chemoradiation (week 6), and at the 6-week follow-up visit. Patients are followed at 1 month, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 244 patients (122 per treatment arm) will be accrued for this study within 38 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed unresectable stage II, IIIA, or IIIB non-small cell lung cancer No distant metastases No prior complete (or gross subtotal) tumor resection No post-resection intrathoracic tumor recurrence Pleural effusion seen on a chest x-ray allowed only if appearing after thoracotomy or other invasive thoracic procedure (pleural effusion acceptable if seen only on CT scan, not on chest x-ray) Must be ineligible or refused participation in protocol RTOG-9309

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Absolute granulocyte count at least 2,000/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 8.0 g/dL Hepatic: Bilirubin no greater than 1.5 mg/dL* SGOT no greater than 1.5 times upper limit of normal* * Unless due to documented benign disease Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No myocardial infarction within the past 6 months No symptomatic heart disease, including angina, congestive heart failure, or uncontrolled arrhythmias Other: No weight loss of greater than 5% in 3 months prior to diagnosis No other prior or concurrent invasive malignancy within the past 3 years except nonmelanomatous skin cancer Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior thoracic or neck radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 1998-09; Primary Completion 2002-07 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Movsas, MD, Study Chair — Fox Chase Cancer Center
Locations (264):
- United States (244):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - Regional Radiation Oncology Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Provena St. Joseph Hospital- Regional Cancer Care Center, Elgin, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - North Mississippi Medical Center/Cancer Center, Tupelo, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Nebraska Health System, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Cooper Cancer Institute, Camden, New Jersey
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fitzgerald Mercy Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Canter Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Machtay M, Bae K, Movsas B, Paulus R, Gore EM, Komaki R, Albain K, Sause WT, Curran WJ. Higher biologically effective dose of radiotherapy is associated with improved outcomes for locally advanced non-small cell lung carcinoma treated with chemoradiation: an analysis of the Radiation Therapy Oncology Group. Int J Radiat Oncol Biol Phys. 2012 Jan 1;82(1):425-34. doi: 10.1016/j.ijrobp.2010.09.004. Epub 2010 Oct 25. PMID 20980108
- [Background] Siddiqui F, Bae K, Langer CJ, Coyne JC, Gamerman V, Komaki R, Choy H, Curran WJ, Watkins-Bruner D, Movsas B. The influence of gender, race, and marital status on survival in lung cancer patients: analysis of Radiation Therapy Oncology Group trials. J Thorac Oncol. 2010 May;5(5):631-9. doi: 10.1097/jto.0b013e3181d5e46a. PMID 20432520
- [Background] Bruner DW. Outcomes research in cancer symptom management trials: the Radiation Therapy Oncology Group (RTOG) conceptual model. J Natl Cancer Inst Monogr. 2007;(37):12-5. doi: 10.1093/jncimonographs/lgm004. PMID 17951225
- [Background] Langer CJ, Swann S, Curran W, et al.: Reassessing prognostic factors in the era of combined modality therapy for locally advanced NSCLC: a retrospective analysis of RTOG 9410 and 9801. [Abstract] Int J Radiat Oncol Biol Phys 63 (2 Suppl 1): A-65, S39, 2005.
- [Background] Machtay M, Swann S, Komaki R, et al.: What is the meaning of local-regional control after chemoradiation for locally advanced NSCLC? An RTOG analysis. [Abstract] Lung Cancer 50 (Suppl 2): A-O-041, S17, 2005.
- [Background] Sause W, Scott C, Byhardt R, et al.: Combined chemotheray radiation therapy treatment in unresected non-small cell lung cancer: Radiation Therapy Oncology Group (RTOG) experience. Lung Cancer 29(suppl 2): 2000.
- [Result] Movsas B, Moughan J, Sarna L, Langer C, Werner-Wasik M, Nicolaou N, Komaki R, Machtay M, Wasserman T, Bruner DW. Quality of life supersedes the classic prognosticators for long-term survival in locally advanced non-small-cell lung cancer: an analysis of RTOG 9801. J Clin Oncol. 2009 Dec 1;27(34):5816-22. doi: 10.1200/JCO.2009.23.7420. Epub 2009 Oct 26. PMID 19858383
- [Result] Sarna L, Swann S, Langer C, Werner-Wasik M, Nicolaou N, Komaki R, Machtay M, Byhardt R, Wasserman T, Movsas B. Clinically meaningful differences in patient-reported outcomes with amifostine in combination with chemoradiation for locally advanced non-small-cell lung cancer: an analysis of RTOG 9801. Int J Radiat Oncol Biol Phys. 2008 Dec 1;72(5):1378-84. doi: 10.1016/j.ijrobp.2008.03.003. Epub 2008 May 22. PMID 18501528
- [Result] Movsas B, Scott C, Langer C, Werner-Wasik M, Nicolaou N, Komaki R, Machtay M, Smith C, Axelrod R, Sarna L, Wasserman T, Byhardt R. Randomized trial of amifostine in locally advanced non-small-cell lung cancer patients receiving chemotherapy and hyperfractionated radiation: radiation therapy oncology group trial 98-01. J Clin Oncol. 2005 Apr 1;23(10):2145-54. doi: 10.1200/JCO.2005.07.167. PMID 15800308
- [Result] Nicolaou N, Moughan J, Sarna L, et al.: Quality of life (QOL) supercedes the classic predictors of survival in locally advanced non-small cell lung cancer (NSCLC): an analysis of Radiation Therapy Oncology Group (RTOG) 9801. [Abstract] Int J Radiat Oncol Biol Phys 69 (3 Suppl): A-103, S58-59, 2007.
- [Result] Sarna L, Swann S, Langer C, et al.: Is there a "disconnect" between physician and patient - reported outcomes (PROs): an analysis of RTOG 98-01. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2595, S541, 2006.
- [Result] Werner-Wasik M, Langer C, Movsas B. Amifostine in chemoradiation therapy for non-small cell lung cancer: review of experience and design of a phase II trial assessing subcutaneous and intravenous bolus administration. Semin Oncol. 2005 Apr;32(2 Suppl 3):S105-8. doi: 10.1053/j.seminoncol.2005.03.018. PMID 16015544
- [Result] Werner-Wasik M, Scott C, Movsas B, et al.: Amifostine as mucosal protectant in patients with locally advanced non-small cell lung cancer (NSCLC) receiving intensive chemotherapy and thoracic radiotherapy (RT): results of the radiation therapy oncology group (RTOG) 98-01 study. [Abstract] Int J Radiat Oncol Biol Phys 57 (2 Suppl): S216, 2003.
- [Result] Movsas B. Exploring the role of the radioprotector amifostine in locally advanced non-small cell lung cancer: Radiation Therapy Oncology Group trial 98-01. Semin Radiat Oncol. 2002 Jan;12(1 Suppl 1):40-5. doi: 10.1053/srao.2002.31362. PMID 11917283
- [Derived] Lawrence YR, Paulus R, Langer C, Werner-Wasik M, Buyyounouski MK, Komaki R, Machtay M, Smith C, Axelrod RS, Wasserman T, Bradley JD, Movsas B. The addition of amifostine to carboplatin and paclitaxel based chemoradiation in locally advanced non-small cell lung cancer: long-term follow-up of Radiation Therapy Oncology Group (RTOG) randomized trial 9801. Lung Cancer. 2013 Jun;80(3):298-305. doi: 10.1016/j.lungcan.2013.02.008. Epub 2013 Mar 7. PMID 23477890